CLINICAL TRIAL: NCT03416660
Title: Comparison Between Effectiveness of Different Densities of Fractional Carbon Dioxide Laser in Treatment of Postburn Scar.
Brief Title: Efficacy of Different Densities of Fractional Carbon Dioxide in Treatment of Post Burn Scars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Suzan Shalaby, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: cairou19
Record Dates: First submitted 2018-01-12; First posted 2018-01-31 (Actual); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Scar
Keywords: Fractional laser; Postburn scar; Density
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Intervention Model Description: The study included 25 Egyptian patients with burn scars recruited from the Out Patient Clinic, Dermatology Department, Cairo University. Each has three post burn scars, assigned to monthly fractional carbon dioxide laser sessions with a total of 3 sessions. parameters are :
  Lesion A or part A parameters: 20 W, 800-1000μs dwell time, 2 to 3 stacks according to scar thickness, 900µm spacing (7.4% density).
  Lesion B or part B parameters: 20 W, 800-1000μs dwell time, 2 to 3 stacks according to scar thickness, 600µm spacing (12.6% density).
  Lesion C or part C parameters: 20 W, 800-1000μs dwell time, 2 to 3 stacks according to scar thickness, 300 µm spacing (25.6% density).
  3 mm punch biopsy is taken before and one month after last session for assessment of collagen via (Masson's trichrome strain). In addition clinical evaluation is done via Vancouver & Patient and Observer Scar Assessment Scale
Who Masked: Outcomes Assessor
Masking Description: masked to the parameters of laser treatment in each lesion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Low density (Active Comparator): Fractional carbon dioxide laser: Lesion A or part A parameters: 20 W, 800-1000μs dwell time, 2 to 3 stacks according to scar thickness, 900µm spacing (7.4% density).
  Interventions: Device: Fractional Carbon Dioxide laser
- Medium density (Active Comparator): Fractional carbon dioxide laser : Lesion B or part B parameters: 20 W, 800-1000μs dwell time, 2 to 3 stacks according to scar thickness, 600µm spacing (12.6% density).
  Interventions: Device: Fractional Carbon Dioxide laser
- High density (Active Comparator): Fractional carbon dioxide laser : Lesion C or part C parameters: 20 W, 800-1000μs dwell time, 2 to 3 stacks according to scar thickness, 300 µm spacing (25.6% density).
  Interventions: Device: Fractional Carbon Dioxide laser

INTERVENTIONS:
Device: Fractional Carbon Dioxide laser

SUMMARY:
This study aims to compare effectiveness of different densities of carbon dioxide fractional laser in the treatment of postburn scar.

DETAILED DESCRIPTION:
The study included 25 Egyptian patients with burn scars recruited from the Out Patient Clinic, Dermatology Department, Cairo University. Each has three post burn scars, assigned to monthly fractional Carbon dioxide laser sessions with a total of 3 sessions. parameters are :

Lesion A or part A parameters: 20 W, 800-1000μs dwell time, 2 to 3 stacks according to scar thickness, 900µm spacing (7.4% density).

Lesion B or part B parameters: 20 W, 800-1000μs dwell time, 2 to 3 stacks according to scar thickness, 600µm spacing (12.6% density).

Lesion C or part C parameters: 20 W, 800-1000μs dwell time, 2 to 3 stacks according to scar thickness, 300 µm spacing (25.6% density).

3 mm punch biopsy is taken before and one month after last session for assessment of collagen via (Masson's trichrome strain). In addition clinical evaluation is done via Vancouver & Patient and Observer Scar Assessment Scale .

ELIGIBILITY:
Inclusion Criteria:

* • Burn scars of at least 1 year duration.

  * Patients with three separate lesions each of them about 2 to 5cm or patients with single lesion equal or more than 8 to 10cm.

Exclusion Criteria:

* • Pregnancy.

  * Lactation.
  * Oral retinoid drugs within the past 6 months.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-23 (Actual)

PRIMARY OUTCOMES:
Clinical improvement Vancouver score | 1 month after last session
  to compare the efficacy of different densities of fractional laser in treatment of post burn scars

CONTACTS AND LOCATIONS:
Overall Officials: SOUZAN M AMIN, Principal Investigator — Cairo University
Locations (1):
- Souzan Mohamed Amin, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No